CLINICAL TRIAL: NCT07123272
Title: Usability of the MeTime MS Acupressure Mobile Application in Adults With MS
Brief Title: Usability of the MeTime MS App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Anna Kratz, Principal Investogator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00268311; K24AT012644 (NIH)
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Pain; Fatigue Symptom
Keywords: chronic pain; acupressure; digital health; fatigue; usability; feasibility
MeSH Terms: conditions — Multiple Sclerosis; Pain; Fatigue; Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxing Self-Acupressure (Experimental): Self-guided use of a smartphone app that informs users how to administer relaxing acupressure each day for 6 weeks.
  Interventions: Behavioral: Self-guided smartphone application for relaxing acupressure
- Stimulating Self-Acupressure (Experimental): Self-guided use of a smartphone app that informs users how to administer relaxing acupressure each day for 6 weeks.
  Interventions: Behavioral: Self-guided smartphone application for stimulating acupressure

INTERVENTIONS:
Behavioral: Self-guided smartphone application for relaxing acupressure — Relaxing Acupressure entails applying pressure with either a finger, pencil, or similar object to acupressure points. For the relaxing protocol, there is a total of 9 acupoints (1 unilateral and 4 bilateral). Each point will be stimulated for 3 minutes, yielding a total treatment time of 27 minutes each day. The acupoints are:
  1. Yin Tang (Unilaterally): Located on the forehead, between the eyebrows.
  2. Anmian (Right and Left/bilaterally): Located on the posterior aspect of the neck, in a slight depression along the bone directly behind the ear.
  3. Heart 7 (HT7) (Right and Left/bilaterally): Located on the palmer surface of the hands on the wrist crease; in line with the pinky.
  4. Spleen 6 (SP6) (Right and Left/bilaterally): Located on the inside of the lower leg, approximately 4 fingers width above the bone of the ankle.
  5. Liver 3 (LIV3) (Right and Left/bilaterally): This point is located on the foot, near the big and second toes.
  Other Names: Me Time MS
  Arms: Relaxing Self-Acupressure
Behavioral: Self-guided smartphone application for stimulating acupressure — There is a total of 10 acupoints (2 unilateral and 4 bilateral). Each point is stimulated for 3 minutes, yielding a total treatment time of 30 minutes each day. The acupoints are:
  1. Du 20 (Unilaterally): Located at the top of the head.
  2. Large Intestine 4 (LI4) (Right and Left/bilaterally): Located on the back of the hand, between your thumb and index finger.
  3. Conception Vessel 6 (CV6) (Unilaterally): Located two finger widths below the navel on the centerline.
  4. Stomach 36 (ST36) (Right and Left/bilaterally): Located on the lower leg below the knee on the outside of the leg.
  5. Spleen 6 (SP6) (Right and Left/bilaterally): Located on the inside of the lower leg, approximately 4 fingers width above the bone of the ankle.
  6. Kidney 3 (K3) (Right and Left/bilaterally): Located on the inside of the ankle.
  Other Names: Me Time MS
  Arms: Stimulating Self-Acupressure

SUMMARY:
The Me Time MS Application was designed to enable self-administration of acupressure. Two forms of acupressure - either "relaxing" or "stimulating" protocols - are administered through the Me Time MS app.

The goal of this study is to assess the usability of the Me Time MS app in a sample of 10 adults with multiple sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* MS diagnosis (all MS subtypes included)
* Age 18 years or older
* Average Fatigue Severity Scale (FSS) score ≥ 4 at screening coupled with the opinion of the volunteer that the fatigue has interfered with their daily activities for ≥ 3 months
* Presence of chronic pain defined as moderate to severe pain for ≥ 3-month duration that is ≥ 4 on average using a 0-10 numerical rating scale
* Home access to internet via Wi-Fi or cellular data
* Active email account

Exclusion Criteria:

* Not fluent in English
* Pregnancy or breast feeding, or anticipate pregnancy in next 6 months
* Inability to use smartphone/tablet and/or MeTime MS mobile app
* Anything at the discretion of the PI or study team that would preclude participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kratz, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
This study's limited qualitative data focused on digital health tool usability is not relevant outside of our efforts to optimize the digital health tool (Me Time MS); therefore release of qualitative data is not planned.

RESULTS

PARTICIPANT FLOW:
Groups:
- Relaxing Self-Acupressure: Self-guided use of a smartphone app that informs users how to administer relaxing acupressure each day for 6 weeks.
  Self-guided smartphone application for relaxing acupressure: Relaxing Acupressure entails applying pressure with either a finger, pencil, or similar object to acupressure points. For the relaxing protocol, there is a total of 9 acupoints (1 unilateral and 4 bilateral). Each point will be stimulated for 3 minutes, yielding a total treatment time of 27 minutes each day. The acupoints are:
  1. Yin Tang (Unilaterally): Located on the forehead, between the eyebrows.
  2. Anmian (Right and Left/bilaterally): Located on the posterior aspect of the neck, in a slight depression along the bone directly behind the ear.
  3. Heart 7 (HT7) (Right and Left/bilaterally): Located on the palmer surface of the hands on the wrist crease; in line with the pinky.
  4. Spleen 6 (SP6) (Right and Left/bilaterally): Located on the inside of the lower leg, approximately 4 fingers width above the bone of the ankle.
  5. Liver 3 (LIV3) (Right and Left/bilaterally): This point is located on the foot, near the big and second toes.
- Stimulating Self-Acupressure: Self-guided use of a smartphone app that informs users how to administer relaxing acupressure each day for 6 weeks.
  Self-guided smartphone application for relaxing acupressure: There is a total of 10 acupoints (2 unilateral and 4 bilateral). Each point is stimulated for 3 minutes, yielding a total treatment time of 30 minutes each day. The acupoints are:
  1. Du 20 (Unilaterally): Located at the top of the head.
  2. Large Intestine 4 (LI4) (Right and Left/bilaterally): Located on the back of the hand, between your thumb and index finger.
  3. Conception Vessel 6 (CV6) (Unilaterally): Located two finger widths below the navel on the centerline.
  4. Stomach 36 (ST36) (Right and Left/bilaterally): Located on the lower leg below the knee on the outside of the leg.
  5. Spleen 6 (SP6) (Right and Left/bilaterally): Located on the inside of the lower leg, approximately 4 fingers width above the bone of the ankle.
  6. Kidney 3 (K3) (Right and Left/bilaterally): Located on the inside of the ankle.
Period: Overall Study
Arm/Group | Relaxing Self-Acupressure | Stimulating Self-Acupressure
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relaxing Self-Acupressure | Stimulating Self-Acupressure | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (7.65) | 54 (9.67) | 51.00 (8.81)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1 | 0 | 1
  Female | 3 | 5 | 8
  Prefer Not to Answer | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10
Education Level [Count of Participants; unit: Participants]
  High school graduate | 1 | 0 | 1
  Associates/Technical Degree | 2 | 1 | 3
  Some college, No Degree | 0 | 1 | 1
  Bachelor's Degree | 1 | 2 | 3
  Master's Degree | 1 | 1 | 2
Employment Status [Count of Participants; unit: Participants]
  Disabled | 3 | 2 | 5
  Working Part time | 0 | 1 | 1
  Working Full Time | 2 | 2 | 4
Multiple sclerosis (MS) Subtype [Count of Participants; unit: Participants]
  Relapsing-Remitting Multiple Sclerosis | 4 | 3 | 7
  Primary Progressive Multiple Sclerosis | 1 | 1 | 2
  Secondary Progressive Multiple Sclerosis | 0 | 1 | 1
Mobility aid [Count of Participants; unit: Participants]
  Walk without assistance | 2 | 2 | 4
  Cane/Walker | 3 | 1 | 4
  Manual Wheelchair | 0 | 1 | 1
  Participant Did Not Respond | 0 | 1 | 1
Patient-determined Disease Steps (PDDS) [Count of Participants; unit: Participants]
  Normal | 1 | 0 | 1
  Mild Disability | 1 | 1 | 2
  Moderate Disability | 0 | 0 | 0
  Gait Disability | 0 | 1 | 1
  Early cane | 2 | 1 | 3
  Late Cane | 1 | 1 | 2
  Bilateral Support | 0 | 0 | 0
  Wheelchair/Scooter | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participant Perception of Me Time MS App Usability
Description: Qualitative descriptions of positive, negative, and neutral aspects of usability of the Me Time MS app, gathered through one-on-one, open-ended interviews after 6 weeks of access to the app. Results reflect the total number of comments across all participants that were provided for each category. Participants could submit multiple types of comments.
Time Frame: Up to 2 weeks after the 6-week app usage period ended
Population: 3 participants in the Stimulating arm did not attend an interview.
Measure: Number; unit: Comments
Units Other Than Participants: Comments
Arm/Group | Relaxing Self-Acupressure | Stimulating Self-Acupressure
Number analyzed (Participants) | 5 | 2
Number analyzed (Comments) | 59 | 21
Comments
  Positive | 37 | 11
  Negative | 9 | 4
  Neutral | 13 | 6

2. Secondary Outcome: System Usability Scale (SUS) Adapted for the MeTime MS App
Description: SUS is a custom, 10-item survey to assess the participant's perception of the usability of the MeTime MS app. Possible total score ranges from 0 (lowest usability) to 40 (highest usability).
Time Frame: Up to 2 weeks after the 6-week app usage period ended
Population: 3 participants in the Stimulating Arm did not complete the SUS survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relaxing Self-Acupressure | Stimulating Self-Acupressure
Number analyzed (Participants) | 5 | 2
score on a scale | 35.8 (2.28) | 29.5 (6.36)

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Arm/Group | Relaxing Self-Acupressure | Stimulating Self-Acupressure
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relaxing Self-Acupressure (N=5) | Stimulating Self-Acupressure (N=5)
Fatigue (General disorders) | 1 | 1
Cramping (Nervous system disorders) | 1 | 0
Soreness (General disorders) | 2 | 0
Difficulty with certain acupoints due to limited mobility (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT07123272/Prot_SAP_001.pdf
  • Informed Consent Form (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT07123272/ICF_000.pdf